CLINICAL TRIAL: NCT00380016
Title: Catheter-Based Treatment of Cardiovascular Disease in Patients
Brief Title: Catheter-Based Treatment of Cardiovascular Disease
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Purpose: Treatment
Other Study IDs: 060203; 06-H-0203
Record Dates: First submitted 2006-09-22; First posted 2006-09-25 (Estimated); Last update posted 2017-07-02 (Actual); Status verified 2009-03-03

CONDITIONS: Obstructive Coronary Artery Disease; Obstructive Peripheral Artery Disease; Structural Heart Disease
Keywords: Angioplasty; Stent; Coronary Artery Disease; Peripheral Artery Disease; Percutaneous Coronary Intervention; CAD; PAD; Cardiovascular Disease
MeSH Terms: conditions — Coronary Artery Disease; Peripheral Arterial Disease; Cardiovascular Diseases | interventions — Angioplasty

INTERVENTIONS:
Procedure: Percutaneous Transluminal Angioplasty

SUMMARY:
This study offers catheter-based treatment of heart or artery disease. This protocol permits treatment of patients with cardiovascular diseases who may not be eligible to participate in current research protocols. The treatment offered in this protocol is not experimental, but rather standard treatment provided in most large referral hospitals in the United States.

Patients 18 years of age and older who are candidates for catheter-based treatment of obstructive artery disease, including blocked blood flow in a coronary artery (artery to the heart) or in an artery of the arm, leg, brain or kidney may be eligible for this study. Candidates are screened with a general medical evaluation that may include blood tests, magnetic resonance imaging, and monitoring of heart rate and rhythm.

Participants undergo angioplasty or stenting for blockage in an artery to the heart or an artery of the arm, leg, brain or kidney. The procedure uses a balloon-tipped catheter to open the blocked artery and likely requires permanent implantation of a metal tube (stent) to improve blood flow through the vessel. During the procedure, the patient is given a sedative and pain medication, if needed.

DETAILED DESCRIPTION:
The NHLBI is developing novel minimally invasive catheter-based treatments for cardiovascular disease. These investigational treatments require that physicians, nurses and technical staff maintain and expand their technical skills in the conduct of conventional catheter-based treatments.

This protocol permits treatment of patients with cardiovascular diseases who are not necessarily eligible to participate in existing clinical research protocols, but who are of medical interest for the purpose of training professional staff, or who may be eligible for adjunctive investigational imaging during clinical treatment. Efforts will be made to offer treatment to patients with limited financial resources or with limited access to specialty health care.

This protocol also provides a mechanism to offer catheter-based treatment of cardiovascular disease to patients, so that they may participate in technical development protocols in cardiovascular intervention or in cardiovascular imaging.

ELIGIBILITY:
* INCLUSION CRITERIA:

Adult men and women with cardiovascular disease will be eligible to participate in this training protocol.

1. Adult men and women, age 18 years or older
2. Eligible for catheter-based treatment. A representative list of diseases and catheter-based treatments includes:

   * Obstructive coronary artery disease manifest as myocardial infarction, angina pectoris, angina-equivalent, ischemic dysrhythmia, or evidence of ischemia or viability on non-invasive cardiovascular testing
   * Obstructive peripheral artery disease manifest as intermittent claudication, limb-threatening ischemia, visceral ischemia, or obstructive extracranial cerebrovascular disease
   * Structural heart disease including patent foramen ovale, atrial septal defect, ventricular septal defect, patent ductus arteriosus, and valvular heart disease

EXCLUSION CRITERIA:

Subjects are excluded if catheter-based therapy is unsuitable, in the opinion of the operating cardiologist.

1. Pregnant women
2. Inability of patient or surrogate to provide informed consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150
Dates: Start 2006-09-20; Study Completion 2009-03-03

CONTACTS AND LOCATIONS:
Locations (1):
- National Heart, Lung and Blood Institute (NHLBI), 9000 Rockville Pike, Bethesda, Maryland, United States